CLINICAL TRIAL: NCT05411055
Title: Aortic Valve Neocuspidization With Glutaraldehyde-Treated Autologous Pericardium
Brief Title: Aortic Valve Neocuspidization With Glutaraldehyde-Treated Autologous Pericardium (Ozaki Procedure)
Acronym: PARACADUTE
Status: Active, not recruiting | Type: Observational
Sponsor: Maria Cecilia Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MCH 2021-02
Record Dates: First submitted 2022-06-06; First posted 2022-06-08 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Aortic Valve Disease
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Ozaki aortic valve reconstruction procedure uses autologous or bovine pericardium as an aortic cusp replacement without the use of struts and with use of the patient's own native aortic root. In this technique one can replace individual aortic cusps, 1, 2, or all 3 cusps. Ideally the patient's autologous pericardium will be harvested and fixed in gluteraldehyde at the time and prepared for the patient's specific annular dimensions with the neoaortic root sizers. Based on the measured size, one then uses a leaflet template to independently replace the cusps resulting in more effective preservation of the natural motion of the aortic valve annulus in coordination of the left ventricle, aortic annulus, sinus of Valsalva, and aorta compared to stented bioprosthetic and/or mechanical aortic valve replacements. Professor Ozaki has now performed 1000 Ozaki neoaortic valve reconstructive operations and has better than 95% freedom from re-operation at late follow-up. The objective of this study is to collect a large collection of prospective data from patients undergoing aortic neocuspidalization surgery for aortic valve insufficiency or stenosis isolated or combined with other procedures

ELIGIBILITY:
Inclusion Criteria:

* severe aortic valve stenosis or insufficiency
* Written informed consent
* Willingness to carry out the follow-up visits

Exclusion Criteria:

* Other types of aortic valve surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing aortic neocuspidal surgery
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-06-06 (Actual); Primary Completion 2026-06-06 (Estimated); Study Completion 2027-06-06 (Estimated)

PRIMARY OUTCOMES:
postoperative complications | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- MCH, Cotignola, Ravenna, Italy